CLINICAL TRIAL: NCT06595940
Title: Genomic Sequencing for Evaluation of Uncommon Disease Manifestations Through the Childhood Complex Disease Genomic Section
Brief Title: Genetic Analysis of Uncommon Disease Presentations in Non-US Populations
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001645; 001645-HG
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-22

CONDITIONS: Undiagnosed Diseases; Rare Diseases
Keywords: Genetics; Genomic sequencing; Under-represented populations; Medical genetics; Clinical Phenotype; Uncommon disease
MeSH Terms: conditions — Undiagnosed Diseases; Rare Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Individuals with a condition that is expected to be caused by a genetic change
- Unaffected: Individuals who are first-degree relatives (parents, siblings, children) of affected individuals enrolled in this study

SUMMARY:
Background:

Genetics research over the past 20 years has helped researchers find the causes of many diseases. More powerful tools for genetic testing now exist. Researchers want to use these new tools to learn more about genetic diseases. They want to look for possible genetic causes of unusual diseases. They will focus on people who live outside of the United States and whose access to genetic testing has been limited.

Objective:

To look for potential genetic sources of diseases among children and their families.

Eligibility:

Children aged 2 to 18 years and their related family members who have or may have a genetic disease. They will reside primarily outside of the US.

Design:

Participants will be recruited at sites outside of the US. Participants will be screened. Their existing medical records will be reviewed. They will have a physical exam. They will answer questions about their family history and symptoms. Participants will provide samples for genetic testing. They may have blood drawn. They may spit saliva into a small container. They may have a cotton swab rubbed on the inside of the mouth. The samples will be shipped to the NIH for genetic testing. Participants will be notified if testing reveals a known disease. Participants may be asked to provide new samples to confirm the diagnosis. Local study teams will contact the participants about the results. Participants will also be notified if analysis yields gene variants that may cause disease.

DETAILED DESCRIPTION:
Study Description:

We plan to couple novel techniques of genomic interrogation with more traditional methods involved in genetic discovery to investigate a broad range of diseases and conditions in locations without access to medical genetics for which there exists strong evidence that genetic factors are contributory.

Objectives:

Primary Objective: To investigate the genetic contribution to conditions displaying unconventional clinical phenotypes/familial segregation among individuals belonging to historically underrepresented populations.

Secondary Objective: To develop an international collaborative network across countries with limited or no access to medical genetics.

Tertiary/Exploratory Objective: To identify the psychosocial impact and cultural considerations of the diagnostic odyssey in countries without medical genetics access to better inform genetic counseling practices for these populations.

Endpoints:

Primary Endpoint: Exhaustion of available genomic interrogation techniques to determine the etiology of unconventional clinical phenotypes.

Secondary Endpoint: Independence and autonomy when conducting genetic studies among sites with limited to no access to medical genetics.

Tertiary/Exploratory Endpoint: Elucidation of psychosocial impact and cultural considerations for patients with limited access to medical genetics.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Probands aged >2 years at enrollment or first-degree relatives of probands (age >2 years).
3. Suspicion of genetic etiology of illness due to strong family history, precocious onset, severity or mildness of phenotype, or all factors being present.
4. Affected individuals and unaffected family members, determination of clinical criteria for inclusion will be determined by medical record review prior to participation.
5. Ability of participant and their parent or guardian to understand and have willingness to sign a written informed consent and/or assent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Anyone unwilling to provide informed consent (for themselves as adults, on behalf of their children as minors, or on behalf of an adult who is unable to provide consent for themselves) or assent.
2. Individuals who have undergone diagnostic testing for a genetic condition AND the test results were positive.
3. Evidence that symptoms are secondary or caused by an undiagnosed condition that is unlikely to have a genetic cause.
4. In the opinion of the investigator, participant has a condition that would preclude participation in the study by interfering with the participant s ability to engage in the required protocol evaluation and testing.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To be eligible to participate in this study, an individual must meet all of the following criteria: willingness to comply with all study procedures and availability for the duration of the study; age >2 years when enrolled in the study; suspicion of genetic cause for illness due to strong family history, young age of onset, illness being either more or less severe than expected; verification of meeting clinical inclusion criteria by reviewing a participant's medical record; ability of participant and their parent or guardian (if <18 years old) to understand and willingly sign informed consent document. Those with previous genetic testing that was positive, those with evidence that their symptoms are caused by a condition unlikely to be genetic, or those with conditions that may interfere with their ability to participate in required testing will be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2034-08-21 (Estimated); Study Completion 2034-08-21 (Estimated)

PRIMARY OUTCOMES:
Exhaustion of available genomic interrogation techniques to determine the etiology of unconventional clinical phenotypes. | 10 years
  The outcome will be achieved when we have reached a point where use of appropriate genomic interrogation techniques does not yield new pathophysiological insights.

SECONDARY OUTCOMES:
Independence and autonomy when conducting genetic studies among sites with limited to no access to medical genetics. | 10 years
  The creation of intra-institutional protocols, relationships with ethics committees, and development of genetic study expertise will indicate this endpoint has been reached.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Hanchard, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- University of Mauritius, Moka, Mauritius

IPD SHARING:
Plan to Share IPD: No